CLINICAL TRIAL: NCT03167853
Title: Phase Ib Study of Safety and Efficacy of Recombinant Humanized Anti-PD-1 Monoclonal Antibody for Patients With Advanced Neuroendocrine Tumors Following Failure of First-Line
Brief Title: Study of JS001 in Patients With Advanced Neuroendocrine Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Principal Investigator, Shen Lin, MD, Professor, Chief of Department of GI Oncology, Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMO-JS001-Ib-NEC-02
Record Dates: First submitted 2017-05-10; First posted 2017-05-30 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- humanized anti-PD-1 monoclonal antibody (Experimental): humanized anti-PD-1 monoclonal antibody is to be injected intravenously 3mg/kg per 2 weeks until disease progresses or unacceptable tolerability occurs.
  Interventions: Biological: humanized anti-PD-1 monoclonal antibody

INTERVENTIONS:
Biological: humanized anti-PD-1 monoclonal antibody — humanized anti-PD-1 monoclonal antibody(JS001) is a programmed death-1 (PD-1) immune checkpoint inhibitor antibody, which selectively interferes with th combination of PD-1 with its ligands, PD-L1 and PD-L2, resulting in the activitation of lymphocytes and elimination of malignancy theoretically.
  Other Names: JS001

SUMMARY:
This is a multi-center, open-label, phase Ib study evaluating safety and efficacy of the humanized anti-PD-1 antibody JS001, as a monotherapy in patients with neuroendocrine tumors who have failed in previous systemic treatment. 40 patients are enrolled and injected with the humanized anti-PD-1 antibody 3mg/mg every 2 weeks until disease progresses or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Must have read, understood, and provided written informed consent voluntarily. Willing to adhere to the study visit schedule and the prohibitions and restrictions specified in this protocol.
2. Male and Female aged 18 and older are eligible;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1;
4. Histologic diagnosis of locally advanced or metastatic nonfunctional neuroendocrine tumors, including well-differentiated neuroendocrine tumors and pooly-differentiated neuroendocrine carcinoma;
5. Ki-67 index ≥10%;
6. Unresectable;
7. Radiographic evidence of disease rogression by RECIST criteria on or after last anti-cancer therapy within 6 months;
8. Prior treatment meeting the following criteria:

   * Patients with pooly-differentiated neuroendocrine carcinomas must have received platinum based lineds of chemotherapy;
   * Patients with well-differentiated neuroendocrine tumors must have received at least one systemic treatment, including somatostatin analogs, mTOR inhibitors, anti-angiogentic agents and chemotherapy;
9. Providing with tumor specimen (for testing the expression of PD L1 and the infiltrating lymphocytes);
10. Predicted survival >=3 months;
11. At least 1 measurable lesion (only 1 measurable lymph node lesion is excluded) (routine CT scan >=20mm, spiral CT scan >=10mm, no prior radiation to measurable lesions);
12. Screening laboratory values must meet the following criteria (within past 14 days): hemoglobin ≥ 9.0 g/dL; neutrophils ≥ 1500 cells/ μL; platelets ≥ 100 x 10^3/ μL; total bilirubin ≤ 1.5 x upper limit of normal (ULN); aspartic transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN without, and ≤ 5 x ULN with hepatic metastasis; serum creatinine ≤1╳ULN, creatinine clearance >50ml/min (CockcroftGault equation) PT/INR, aPTT≤1.5 x ULN;
13. Without systemic steroids within past 4 weeks;
14. Brain or meningeal metastases must be disposed with surgery or radiation, and be stable clinically for at least 3 months (prior systemic steroids was allowed, but concurrent administration of systemic steroids with the study drug is excluded);
15. Males or female of childbearing potential must: agree to use using a reliable form of contraception (eg, oral contraceptives, intrauterine device, control sex desire, double barrier method of condom and spermicidal) during the treatment period and for at least 12 months after the last dose of study drug.

Exclusion Criteria:

1. Prior treatment with antiPD1/PDL1/PDL2 antibody;
2. Hypersensitivity to recombinant humanized antiPD1 monoclonal Ab or its components;
3. Prior treatment with mAb within past 4 weeks;
4. Prior antitumor therapy (including corticosteroids and immunotherapy) or participation in other clinical trials within past 4 weeks, or have not recovered from toxicities since the last treatment;
5. Pregnant or nursing;
6. Positive tests for HIV, HCV, HBsAg or HBcAb with positive test for HBV DNA (>500IU/ml);
7. History with tuberculosis;
8. Patients with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, such as hypophysitis, pneumonia, colitis, hepatitis, nephritis, hyperthyroidism or hypothyroidism;
9. Severe, uncontrolled medical condition that would affect patients' compliance or obscure the interpretation of toxicity determination or adverse events, including active severe infection, uncontrolled diabetes, angiocardiopathy (heart failure > class II NYHA, heart block >II grade, myocardial infarction, unstable arrhythmia or unstable angina within past 6 months, cerebral infarction within past 3 months) or pulmonary disease ( interstitial pneumonia, obstructive pulmonary disease or symptomatic bronchospasm);
10. Evidence with active CNS disease;
11. Meningeal carcinomatosis;
12. Prior treatment with bone marrow stimulating factors，such as CSF (colony stimulating factor), EPO (erythropoietin), within past 2 weeks;
13. Prior live vaccine therapy within past 4 weeks;
14. Prior major surgery within past 4 weeks (diagnostic surgery excluded);
15. Psychiatric medicines abuse without withdrawal, or history of psychiatric illness;
16. Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal cell skin cancer or carcinoma in situ of the cervix;
17. Underlying medical condition that, in the Investigator's opinion, would increase the risks of study drug administration or obscure the interpretation of toxicity determination or adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2019-05-11 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  CT/MRI will be performed every 2 cycles of treatment by RECIST 1.1(each cycle is 21 days))

SECONDARY OUTCOMES:
Duration of response (DOR) | baseline, every 8 weeks up to 1 year after last patient first treatment
  Duration of Response by irRC and RECIST 1.1
Progression-free survival | baseline, every 8 weeks up to 1 year after last patient first treatment
  Progression-free survival is defined as the time from the date of first dose to the date of the first documented radiological progression or death due to any cause
Overall survival | Every 3 months after last visit up to 2 year after last patient first treatment
  Overall survival is defined as the time from date of start of treatment to date of death due to any cause
Immune Response Criteria by irRECIST (immune response duration of response) | baseline, every 8 weeks up to 1 year after last patient first treatment
  Immune Response Criteria by irRECIST and as per BIRC (immune response duration of response)
Immune Response Criteria by irRECIST (immune response overall response rate) | baseline, every 8 weeks up to 1 year after last patient first treatment
  Immune Response Criteria by irRECIST and as per BIRC (immune response overall response rate)
Biochemical response | baseline, 6th week, 16th week
  Changes from baseline in chromogranin-A
Correlation analysis of PD-L1/CD8 expression of tumor and ORR | 3 years
  Changes from baseline in PD-L1/CD8 expression
Correlation analysis of circulating tumor cells (CTC) and ORR | baseline, 8th week
  Changes from baseline of circulating tumor cells (CTC)

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, PhD, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu M, Zhang P, Zhang Y, Li Z, Gong J, Li J, Li J, Li Y, Zhang X, Lu Z, Wang X, Zhou J, Peng Z, Wang W, Feng H, Wu H, Yao S, Shen L. Efficacy, Safety, and Biomarkers of Toripalimab in Patients with Recurrent or Metastatic Neuroendocrine Neoplasms: A Multiple-Center Phase Ib Trial. Clin Cancer Res. 2020 May 15;26(10):2337-2345. doi: 10.1158/1078-0432.CCR-19-4000. Epub 2020 Feb 21. PMID 32086343